CLINICAL TRIAL: NCT06818292
Title: Investigation of the Relationship Between Peripheral and Central Metabolic Changes Induced by GLP-1 Agonists
Acronym: GLPsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nils Opel (Other)
Collaborators: University Hospital, Bonn (Other); Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Sponsor-Investigator, Nils Opel, Prof Dr med, Jena University Hospital
Organization: Jena University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2024-3513-BO
Record Dates: First submitted 2025-01-17; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: GLP-1; MR Spectroscopy; fMRI; Metabolism
MeSH Terms: interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GLP-1 then Placebo (Experimental): Participants will be randomly assigned to receive equivalent volumes of either Placebo (NaCl) or 0.6 mg of the pre-filled solutions from pen-injector Liraglutide (GLP-1 Agonist) in a randomized, counterbalanced order. The administration will occur at two time points: T1 and T3 with a washout period of at least 1 day between the two interventions to minimize carryover effects.
  Interventions: Biological: Liraglutide; Biological: Placebo
- Placebo then GLP-1 (Experimental): Participants will be randomly assigned to receive equivalent volumes of either Placebo (NaCl) or 0.6 mg of the pre-filled solutions from pen-injector Liraglutide (GLP-1 Agonist) in a randomized, counterbalanced order. The administration will occur at two time points: T1 and T3 with a washout period of at least 1 day between the two interventions to minimize carryover effects.
  Interventions: Biological: Liraglutide; Biological: Placebo

INTERVENTIONS:
Biological: Liraglutide — 0.6 mg of the pre-filled solutions from pen-injector Liraglutide (GLP-1 Agonist)
  Other Names: GLP-1 Agonist
Biological: Placebo — 0.1 mL NaCl

SUMMARY:
This study aims to investigate the acute effects of Liraglutide, a GLP-1 receptor agonist established in the treatment of type 2 diabetes and obesity, on brain metabolism, brain network function, and executive functioning as well as mood in healthy, normal-weight individuals. Given the emerging evidence of GLP-1's impact on brain function, including the modulation of reward processing and cognitive functions, this study will focus on the physiological changes induced by Liraglutide and their potential implications for brain health. The overall goal of this study is to assess how acute GLP-1 administration influences systemic and brain metabolism to modulate brain signalling and behaviour.

DETAILED DESCRIPTION:
Glucagon-like Peptide 1 (GLP-1) is a hormone secreted primarily by intestinal epithelial cells that plays a central role in promoting insulin secretion and reducing hunger and food intake. Liraglutide, a GLP-1 receptor agonist, has established benefits in regulating blood glucose and appetite and also directly acts on the brain through GLP-1 receptors. These receptors are widely distributed across brain regions, with high densities in the hypothalamus, brain stem, hippocampus, and in reward-related areas such as the ventral tegmental area (VTA) and nucleus accumbens (NAc). However, the underlying effects of GLP-1 receptor activation on brain metabolism and functional brain networks remain poorly understood.

This study will address several key questions regarding the molecular, cellular, and cognitive changes that occur following the acute administration of Liraglutide. In particular, the investigation will focus on how GLP-1 administration modulates peripheral and central metabolism and on the influence of changes in brain metabolism on signaling. Furthermore, the relationship between brain metabolism, signaling, and psychological as well as cognitive outcomes will be examined.

Magnet resonance spectroscopy (MRS) will be used to measure changes in brain metabolism, with a focus on alterations in key metabolic pathways involved in neuronal function and energy homeostasis. In addition, biochemical profiles in blood will be examined to assess how peripheral metabolic changes may reflect or influence brain metabolism. Functional magnetic resonance imaging (fMRI) will also be employed to determine whether the observed alterations in brain metabolism correlate with changes in brain network connectivity and activity. Finally, correlations between these metabolic and connectivity changes and improvements in cognitive function and psychological parameters, such as executive function and mood (compared to placebo), will be evaluated.

The expected outcomes of this study are important insights into the neurobiological effects of Liraglutide and its potential to influence brain metabolism and functional dynamics. By elucidating the impact of GLP-1 analogues on brain metabolism and cognitive function, a better understanding of how metabolic regulation can affect brain signaling is anticipated. Given the prevalence of cognitive deficits in various psychiatric and neurological conditions, including obesity and type 2 diabetes, this research has the potential to contribute to the development of future therapeutic strategies involving GLP-1 receptor agonists.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight at study inclusion (BMI 18.5-25)
* Generally good physical condition without serious previous illnesses

Exclusion Criteria:

* MRI contraindication: cardiac pacemakers, hearing aids, neurostimulation, insulin pumps, other potentially ferromagnetic implants, screws, clips, prostheses, metal splinters, etc., pregnancy, claustrophobia, extensive tattoos, medication that impairs thermoregulation
* Comorbidity: neurological or psychiatric conditions, cognitive impairments, chronic somatic disorders
* Intake of more than 40g of pure alcohol (for men) or more than 20g of pure alcohol (for women), smoking, regular drug use
* Pregnancy or nursing
* Current or within the past five years eating disorder, vegan diet or fasting within the past six months
* Regular medication intake
* Liraglutide contraindications: Hypersensitivity to liraglutide or other components of the medication, medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia endocrine neoplasia syndrome type 2 (MEN2) in personal or family history, history of pancreatitis, current pregnancy or breastfeeding, severe gastrointestinal motility disorders including gastroparesis, severe or terminal renal insufficiency

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Neuropsychology: Processing speed | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  Number Symbol Test, Letter-Number-Symbol Test, TMT-A. A composite score for processing speed will be derived from the Number Symbol Test, Letter-Number Symbol Test, and TMT-A. First, raw scores from each test will be normalized (e.g., converted into z-scores), taking into account that lower completion times on the TMT-A indicate better performance. The normalized scores will then be combined-after adjusting the direction of scores if necessary-by calculating their average to yield a single, unified measure of processing speed.
Neuropsychology: Attention | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  TMT-B, D2-Test. A composite attention score will be created using the D2-Test and TMT-B. Raw scores from both tests will be standardized (e.g., as z-scores). For tests such as the TMT-B, if necessary, the scores will be adjusted (e.g., reverse-coded) so that higher values indicate better attention performance. The resulting standardized scores will be averaged to form a unified attention measure.
Neuropsychology: Memory | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  VLMT-A, block span. A composite memory score will be computed from the VLM-T and Block Span test. Raw scores from each test will be standardized (e.g., into z-scores). These z-scores will then be averaged to yield a single measure of memory performance, reflecting both verbal and visuospatial working memory components.
Neuropsychology: Verbal Fluency | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  MWT-B, Regensburg Word Fluency Test. A composite score for verbal fluency will be derived from the Regensburg Word Fluency Test and the MWT-B. First, raw scores for each test will be converted to standardized scores (e.g., z-scores). If needed, scores will be adjusted so that higher values consistently represent better performance. The standardized scores will then be averaged to create a single composite measure of verbal fluency.
MR spectroscopy | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  metabolites between 0-4 ppm in the posterior cingulate cortex (PCC), medial cingulate cortex (MCC), and anterior insula
Exploratory Proteomics of Autophagy Processes I | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  protein levels of autophagy biomarkers (e.g. LC3II & p62) of isolated PBMCs (peripheral blood mononuclear cells) by Western Blotting
Exploratory Proteomics of Autophagy Processes II | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  protein levels and protein phosphorylation by targeted and untargeted mass spectrometry-based proteomics and phosphoproteomics of isolated PBMCs (peripheral blood mononuclear cells)

SECONDARY OUTCOMES:
Functional MRI | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  resting state connectivity
Structural MR imaging | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  cortical thickness, grey matter volume
Sleep | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  Pittsburgh Sleep Quality Index (PSQI). The 19 self-rated questions of the PSQI are grouped into 7 components. Each component is scored from 0 to 3 points. The scores of the 7 components are then summed to yield a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality.
Depression | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  Beck's depression inventory (BDI-II). The questionnaire consists of 21 questions. Each question is scored on a 4-point scale ranging from no impairment (0) to severe impairment (3). The maximum score is 63.
Anxiety | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  State-Anxiety Inventory (STAI-S). For the STAI-S assessment, specific items (1, 2, 5, 8, 10, 11, 15, 16, 19, and 20) were reverse-coded because they represent aspects of anxiety expressed in a negative direction. After recoding, responses for all STAI-S items were summed to obtain the final test score for state anxiety.
Anhedonia | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  Snaith-Hamilton-Pleasure-Scale (SHAPS). For scoring, each non-affirmative response ("does not apply" or "does not apply at all") is assigned 1 point, while each affirmative response is assigned 0 points. The points are summed across all items, resulting in a total score ranging from 0 to 14, with higher scores indicating a greater degree of anhedonia.
Life quality | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  Positive Mental Health Scale. 9 items rated on a 4-point Likert scale ranging from 0 ("do not agree") to 3 ("completely agree"). A total score is computed by summing the responses to all items, with higher scores indicating greater positive mental health.
Numeric Analog Scales | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  Assessing mood on 0-10 points and sleep duration on 0-13 points scale
Fatigue | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  Fatigue Assessment Scale (FAS), 10-item self-assessment scale. For scoring, responses to items 1-3 and 5-9 are rated on a scale from 1 to 5, while items 4 and 10 are reverse-coded (scored from 5 to 1). The scores for all items are then summed to produce the total FAS score.
Metabolic processes | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  Targeted and quantitative analysis by mass spectrometry
Lipid profiling | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  Targeted and quantitative analysis by mass spectrometry
Transcription expression patterns | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  Gene expression profile by RNA sequencing of isolated PBMCs (peripheral blood mononuclear cells)
Proteome/phosphoproteome/ubiquitinome patterns | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  proteome expression patterns through blood based proteome, phosphoproteome, and ubiquitinome analysis
Exosomal protein patterns | Outcome measures are assessed during a one-week on-site visit per participant (placebo vs. liraglutide days) within an overall study period of 2 months
  Evaluate exosomal protein content through blood based metabolome analysis

CONTACTS AND LOCATIONS:
Overall Officials: Sharmili Edwin Thanarajah, PD Dr med, Principal Investigator — Goethe University; Nils Gassen, Prof Dr, Principal Investigator — University Hospital, Bonn
Locations (1):
- Department of Psychiatry and Psychotherapy, University Hospital Jena, Jena, Thuringia, Germany